CLINICAL TRIAL: NCT02167022
Title: Intense Physiotherapies to Improve Function in Young Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Tucson Medical Center (Unknown); Phoenix Children's Hospital (Other); United Cerebral Palsy-Central Arizona (Unknown); Nemours Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1401195212; 1R01HD079498-01 (NIH)
Record Dates: First submitted 2014-06-12; First posted 2014-06-18 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy
Keywords: intense therapy; brain plasticity; Perception-Action approach
MeSH Terms: conditions — Cerebral Palsy | interventions — Restraint, Physical; Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intense Physiotherapy (Group 1) (Experimental): 30 minutes each of physical and occupational therapy each weekday for 12 weeks (intense physiotherapy) followed by the same therapies administered once a week for 36 weeks (the current standard of care).
  Interventions: Other: Physical and occupational therapy
- Delayed Intense Physiotherapy (Group 2) (Experimental): 30 minutes each of physical and occupational therapy once a week for 36 weeks (the current standard of care) followed by the same therapies administered each weekday for 12 weeks (intense physiotherapy).
  Interventions: Other: Physical and occupational therapy

INTERVENTIONS:
Other: Physical and occupational therapy — The type of physiotherapy to be administered is Perception-Action (P-A). The P-A (motor) intervention is a child-driven approach without the need for special equipment and considers the child and environment as a single unit.Treatment is a coupling of the child with the environment. The environment is changed to enable, enhance or stimulate movement. The action is initiated by the child with the therapist augmenting the child's environment using touch (tactile information) or light support (cushions, bolsters, and gentle touch or pressure) to assist and/or alter the child's active movement. Toys are used and positioned in different places to encourage movement of upper and lower extremities and the trunk; reaching, turning, sitting balance, crawling, walking.

SUMMARY:
Cerebral palsy (CP) is a non-progressive disorder caused by an insult or injury to the brain when the brain is most rapidly developing and which results in some motor dysfunction. Causes for the injury to the brain are numerous and can occur prior to birth, during the birth process, or within the first few months following birth. The motor dysfunction can involve any or all four extremities but most often affects the legs, causing abnormal ambulation. The level of severity depends on the extent of the injury to the brain and can be mild to severe. In severe instances, the child is dependent on others for all his/her care.

There is no known cure for CP, but physical and occupational therapies are administered in an attempt to improve function. The frequency of these therapies varies from once a week (the standard of care in the Western Hemisphere) to five times a week (the standard of care in Asia and some Eastern European countries). The current understanding of brain plasticity offers a theoretical explanation to justify the more intense approach. Active repetitive motor skill-directed rehabilitation utilizes the plasticity of the brain and can restore some function. Intense active physiotherapy can stimulate non-injured but 'dormant' neurons and prevent their 'natural' degeneration in order for them to substitute for the function of injured neurons. It is the very young brain that is most likely to respond to this therapy.

The aim of this proposal is to evaluate the effect of administering both physical and occupational therapy five times each week for 12 weeks and compare it with the standard of care (SOC) approach of one time each week in children between the ages of 12 months and 36 months. This is the first randomized crossover trial to both enroll this young a population of children with cerebral palsy as well as to evaluate this approach from both the therapists and the parents perspectives. The number of children that this study will enroll is larger than in most CP studies. The children will be evaluated clinically with two validated instruments, one of which was designed specifically for children with CP and is administered and scored by certified therapists and the other which was designed for children with developmental disabilities and is scored by the child's care provider. A sub-set of children will have a special type of MRI to evaluate any changes in the neurological structure of the brain.

The Department of Pediatrics at the University of Arizona recently completed a collaborative study with the Neurologic Department at the Beijing Children's Hospital where the intense approach of five therapies per week is the SOC. The positive results prompted another investigation to determine if such an approach would be feasible in the United States. A compliance rate of 81% confirmed feasibility and the perception that parents who have a child diagnosed with CP will do whatever they can to improve their child's motor function.

DETAILED DESCRIPTION:
Specific Aim #1: To compare the effectiveness of an intense physiotherapy program with the current standard of care in the management of children with spastic cerebral palsy.

Hypothesis #1: Children receiving a short cluster of intense therapies (5 times per week for 12 weeks) will show greater functional gains as determined by the Gross Motor Function Measure (GMFM-66) and the Pediatric Evaluation Disability Inventory (PEDI) than those receiving the same therapies once a week, the current standard of care.

Specific Aim #2: To determine if the functional gains by children with spastic cerebral palsy achieved with an intense physiotherapy program will continue to improve while receiving less intense standard weekly therapies for at least 36 weeks (9 months) following completion of the intense program.

Hypothesis #2: Motor skills gained after 12 weeks of intensely administered physiotherapies as determined by the GMFM and the PEDI will continue to improve at a rate greater than that seen in children receiving the same therapies once a week, the current standard of care.

Specific Aim #3: After receiving the same number of therapies at the end of the 48-week protocol, children receiving the intense series of therapies during the first 12-weeks will have made greater functional gains than those receiving them during the last 12-weeks.

Hypothesis #3: Children who receive intense physiotherapies at an earlier age make greater gains then those who receive the same therapies at a later age.

Specific Aim #4: To develop a clinical profile that will identify those children most likely to benefit from intensely administered physiotherapies.

Hypothesis #4: Clinical and radiologic characteristics play a major role in response to therapy.

Explorative Aim: To assess the correlation between clinical improvement from intense physiotherapies and anatomical changes using magnetic resonance imaging (MRI).

Hypothesis: The improvements from intense physiotherapies seen in the clinical assessments will be reflected by alterations of brain connectivity parameters available from neuroanatomical MRI and diffusion tensor imaging (DTI).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 12 to 36 months of age (The diagnosis of CP is often uncertain under the age of 12 months. The cutoff at 36 months is to have a population of young children when the brain is most "plastic" and most susceptible to reorganization).
2. Diagnosis: Diagnosis of spastic CP confirmed by a pediatric neurologist or pediatric rehabilitation specialist.
3. Etiology: The insult to the central nervous system that caused the motor dysfunction must have occurred during gestation or within one year after birth independent of gestational age.
4. Disease severity level: Gross Motor Function Classification System (GMFCS) levels I, II and III.

Exclusion Criteria:

1. Diagnosis: Diagnosis of CP secondary to neuronal migration.
2. Co-morbidities: Medical conditions that may prevent the administration of rehabilitation therapies at the intensity required by the study, or that may compromise the study ability to maintain blindness, or that have a co-morbidity not typically associated with CP (i.e. cancer, cystic fibrosis).
3. Co-interventions: Anticipated pharmacological intervention or procedure or participation in other studies that may interfere with this study.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure-66 (GMFM-66) | Change from Baseline at 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  The primary aim is to assess function. The evaluation instruments we chose are standard in CP research and include an assessment by a certified therapist of Gross Motor Function Measure-66 (GMFM-66) and a parental assessment of the child's functional abilities in the home environment (PEDI-FS). For the primary and secondary outcomes, these endpoints will be assessed at baseline and at 12 weeks as well as every 12 weeks for the next 36 weeks. The evaluation at 48 weeks after the completion of the intense schedule allows an estimation of the persistence of change.
  The GMFM-66 is a criterion referenced validated instrument that has been shown to detect change in gross motor function (performance) of children with CP as a result of various interventions. The 66 test items have been grouped into five dimensions: (1) lying and rolling; (2) crawling and kneeling; (3) sitting, standing and walking; (4) running, and (5) jumping.

SECONDARY OUTCOMES:
Change in Pediatric Evaluation of Disability Inventory-Functional Skills (PEDI-FS) | Change from Baseline at 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  The primary aim is to assess function. The evaluation instruments we chose are standard in CP research and include an assessment by a certified therapist of Gross Motor Function Measure-66 (GMFM-66) and a parental assessment of the child's functional abilities in the home environment (PEDI-FS). For the primary and secondary outcomes, these endpoints will be assessed at baseline and at 12 weeks as well as every 12 weeks for the next 36 weeks. The evaluation at 48 weeks after the completion of the intense schedule allows an estimation of the persistence of change.
  The PEDI-FS is an instrument developed specifically for children from 6 months through 7 years of age who have some type of a disability. It is a child's primary care provider's assessment of what skills the child is able to perform. The skills are grouped into three domains: (1) self-care, (2) mobility, and (3) social function.

OTHER OUTCOMES:
Change in Magnetic Resonance Imaging (MRI)/Diffusion Tensor MRI (DTI) | Change from Baseline at 36 weeks
  As part of an exploratory aim, imaging studies will be done at the Barrow Neurological Institute at Phoenix Children's Hospital on a small subset of enrolled children with hemiplegia. Ten children from each of the two randomized groups stratified for age and severity will be imaged before therapy and at 36 weeks after the beginning of therapy. The purpose of this subset is to evaluate white matter integrity and connectivity throughout the entire brain. Differences at 36 weeks will be indicative of alterations in white matter and connectivity scores due to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Burris R Duncan, MD, Principal Investigator — University of Arizona
Locations (4):
- United States (4):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - United Cerebral Palsy-Central Arizona, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Nemours Children's Hospital, Orlando, Florida